CLINICAL TRIAL: NCT06266871
Title: SOX Combined With Tislelizumab and Low-dose Radiation Therapy for Neoadjuvant Treatment of Locally Advanced Gastric/Gastroesophageal Junction Adenocarcinoma: a Prospective, Multi-center, Single-arm, Phase Ib/II Clinical Trial
Brief Title: SOX Combined With Tislelizumab and LDRT for Neoadjuvant Treatment of Locally Advanced Gastric Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ming Liu, Clinical Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WCH-2023-1625
Record Dates: First submitted 2024-01-31; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SOX+Tislelizumab+LDRT (Experimental): Laparoscopic exploration is required in all patients to detect occult peritoneal metastases.
  All patients will start with one cycle of neoadjuvant therapy of SOX plus tislelizumab regimen: S-1: 40-60 mg Bid, d1-14, q3w; oxaliplatin: 130 mg/m2, iv drip, d1, q3w; tislelizumab: 200 mg, iv drip, d1, q3w.
  Then, LDRT will be performed in the target area (including the primary gastric lesion and positive/suspected positive lymph nodes).
  After radiotherapy, patients will receive another two cycles of SOX plus tislelizumab regimen.
  Radical D2 gastric cancer resection will be performed 4-6 weeks after the last administration of SOX plus tislelizumab regimen.
  The adjuvant therapy will start in 4-6 weeks after the surgery, and we recommend adjuvant treatment with SOX regimen for up to 5 cycles.
  Interventions: Drug: SOX+Tislelizumab+LDRT

INTERVENTIONS:
Drug: SOX+Tislelizumab+LDRT — All patients will start with one cycle of neoadjuvant therapy of SOX plus tislelizumab regimen: S-1: 40-60 mg Bid, d1-14, q3w; oxaliplatin: 130 mg/m2, iv drip, d1, q3w; tislelizumab: 200 mg, iv drip, d1, q3w.
  LDRT will be performed in the target area. After radiotherapy, patients will receive another two cycles of SOX plus tislelizumab.
  Radical D2 gastric cancer resection will be performed 4-6 weeks after the last administration of SOX plus tislelizumab.
  The adjuvant therapy will start in 4-6 weeks after the surgery, and we recommend adjuvant treatment with SOX regimen for up to 5 cycles.

SUMMARY:
Neoadjuvant chemotherapy or chemoradiotherapy has become the standard neoadjuvant regimen for locally advanced G/GEJ cancer and has been recommended by a series of treatment guidelines. Although with clinical benefits of neoadjuvant chemotherapy or chemoradiotherapy, the pCR and long-term survival rates are still unsatisfactory and perioperative treatment mode for locally advanced G/GEJ cancer still needs further optimization. In this study, we will explore the efficacy and safety of chemotherapy combined with tislelizumab and LDRT in the neoadjuvant treatment for locally advanced G/GEJ cancer.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm, phase Ib/II trial. In the phase Ib, 5 cases will be enrolled in each treatment group. In the phase II study, a total of 44 patients will be enrolled. Eligible patients will be registered and receive three cycles of SOX plus tislelizumab regimen. Simultaneously, LDRT will be planned and administered. Radical D2 gastric cancer resection will be performed 4-6 weeks after the last administration of chemotherapy plus tislelizumab. The primary endpoint of Phase Ib is to determine the optimal radiation dose for phase II study. The primary endpoint of phase II is the pathological complete response (pCR) rate. Secondary endpoints include R0 resection rate, major pathological response (MPR), objective response rate (ORR), 2-year disease-free survival (DFS) rate, 2-year overall survival (OS) rate and safety profile of the neoadjuvant regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. Histologically or cytologically confirmed diagnosis of locally advanced G/GEJ adenocarcinoma (cT3-T4a, N+, M0) as assessed by exploratory laparoscopic surgery, ultrasonography and/or CT/MRI.
3. Resectable G/GEJ cancer, as judged by experienced surgeons.
4. Eastern Cooperative Oncology Group performance score (ECOG PS) ≤1.
5. Agree to provide blood, feces, and tissue specimens.
6. The expected survival is longer than 3 months.
7. There was no previous antitumor treatment (including chemotherapy, radiotherapy, targeted therapy, immunotherapy, interventional therapy, and other treatments with antitumor effects).
8. Adequate organ and hematological function.
9. Strict contraception.
10. Patients must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.

Exclusion Criteria:

1. Undergoing other drug clinical trials or having participated in any drug clinical trials one month before enrollment.
2. Other tumors that have not been treated or exist at the same time, except carcinoma in situ of the cervix, treated basal cell carcinoma or superficial bladder tumor. If the tumor was cured and no evidence of disease was found for more than 3 years, the patient can be enrolled. All other tumors must be treated at least 3 years before enrollment.
3. Allergic to oxaliplatin, S-1, tislelizumab and similar drugs, or suspected allergies.
4. With serious gastrointestinal diseases that affect the absorption of oral chemotherapy drugs, such as chronic inflammatory bowel disease.
5. History of gastric perforation within 6 months.
6. Clinical manifestations include significant arrhythmia, myocardial ischemia, severe atrioventricular block, heart failure, and severe heart valve disease; Or those with severe lung function impairment; Or those with impaired blood system, liver and kidney function who cannot tolerate radiotherapy and chemotherapy; Or severe bone marrow failure; Or those with uncontrollable infections.
7. With uncontrollable mental illness.
8. Pregnant or lactating women.
9. Unable to comply with the research program or procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-03-10 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
pCR rate | 5 months after the last subject participating in
  defined as the absence of viable tumor cells assessed by histological evaluation criteria after neoadjuvant therapy

SECONDARY OUTCOMES:
R0 resection rate | 5 months after the last subject participating in
  defined as the rate of the complete surgical removal of any residual cancer cells in the tumor bed
MPR rate | 5 months after the last subject participating in
  defined as tumor residual cells ≤10% in the surgical specimen
ORR | 5 months after the last subject participating in
  defined as the proportion of patients with the best overall response of complete response (CR) or partial response (PR)) before surgery
2-year disease-free survival (DFS) rate | every 3 month postoperation up to 24 months
  defined as the proportion of patients without disease relapse 2 years after enrolment
2-year OS rate | every 3 month postoperation up to 24 months
  defined as the proportion of patients survived 2 years after enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Mojin Wang, M.D., Study Director — West China Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang PF, Chen Y, Li WK, Luo ZM, Chen J, Qian K, Chen XD, Wang MJ, Liu M. SOX combined with tislelizumab and low-dose radiation therapy for the neoadjuvant treatment of locally advanced gastric/gastroesophageal junction adenocarcinoma: study protocol for a prospective, multicenter, single-arm, phase Ib/II clinical trial. Front Immunol. 2024 Nov 13;15:1431957. doi: 10.3389/fimmu.2024.1431957. eCollection 2024. PMID 39606219